CLINICAL TRIAL: NCT04857502
Title: 99mTc-PSMA-I&Amp;S in Patients With Prostate Cancer: An Exploratory Biodistribution Study With Histopathology Validation
Brief Title: 99mTc-PSMA-I&S Biodistribution in Patients With Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-002256; NCI-2021-01793 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-01; First posted 2021-04-23 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-01

CONDITIONS: Prostate Carcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (99mTc-PSMA-I&S, SPECT/CT) (Experimental): The first 5 patients receive an initial dose of undergo 99mTc-PSMA-I&S IV followed by 5 SPECT/CT scans at 3-5, 5-20, 17-21, 25-29, and 40-46 hours later. These 5 patients then receive a second dose of 99mTc-PSMA-I&S IV and then undergo standard of care surgery. All subsequent patients receive one dose of 99mTc-PSMA-I&S IV before standard of care surgery.
  Interventions: Drug: 99mTc-based PSMA Imaging and Surgery Agent; Procedure: Computed Tomography; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Drug: 99mTc-based PSMA Imaging and Surgery Agent — Given via IV injection
Procedure: Computed Tomography — Undergo SPECT/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This exploratory study conducted under the RDRC program studies the biodistribution of 99mTc-PSMA-I&S in patients with prostate cancer who undergo pelvic lymph node dissection. Prostate specific membrane antigen (PSMA)-targeted radio-guided surgery uses the preoperative intravenous administration of a PSMA-ligand called PSMA-imaging and surgery (I&S) labeled with the gamma-emitter radioisotope Technetium-99m (99mTc). Giving 99mTc-PSMA-I&S may detect PSMA-expressing lymph nodes during surgery using a gamma probe and may help guide doctors to detect prostate cancer that has spread to the lymph nodes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the biodistribution of 99mTc-based PSMA imaging and surgery agent (99mTc-PSMA-I&S) in normal and malignant tissues of patients with prostate cancer (PCa) with histopathology validation, when available.

SECONDARY OBJECTIVES:

I. To correlate the 99mTc-PSMA-I&S accumulation within tumor lesions observed by in-vivo single-photon emission computed tomography (SPECT), ex-vivo gamma measurements and level of prostate-specific membrane antigen (PSMA) expression quantified by histopathology, when available.

II. To define the best time-point for radio-guided surgery (RGS) with the highest tumor-to-background ratio following 99mTc-PSMA-I&S administration.

OUTLINE:

The first 5 patients receive an initial dose of 99mTc-PSMA-I&S intravenously (IV) followed by 5 SPECT/CT scans at 3-5, 5-20, 17-21, 25-29, and 40-46 hours later. These 5 patients then receive a second dose of 99mTc-PSMA-I&S IV and then undergo standard of care surgery. All subsequent patients receive one dose of 99mTc-PSMA-I&S IV before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men with PCa (primary or recurrent disease)
* Men who received a 68Ga-PSMA-11 positron emission tomography (PET)/computed tomography (CT) for staging or restaging
* Men with evidence of lymph nodes (LNs)-positive disease on 68Ga-PSMA-11 PET/CT
* Men who are scheduled for pelvic LN dissection (PLND)
* Men who can provide oral and written informed consent
* Men who can comply with study procedures

Exclusion Criteria:

* Patients who started any PCa treatment between study enrollment and surgery
* Technically inaccessible nodal location

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The biodistribution of 99mTc-PSMA-I&S in normal and malignant tissues of patients with prostate cancer will be measured by average and maximum standardized uptake value (SUVmean and SUVmax) | time from injection to imaging (range: 1-46 hours)

SECONDARY OUTCOMES:
99mTc-PSMA-I&S accumulation within tumor lesions observed by in-vivo SPECT (SUVmean and SUVmax) will be correlated with ex-vivo gamma measurements (counts/minute) and level of PSMA expression quantified by histopathology (IHC score) | time from injection to imaging (range: 1-46 hours)
The best time-point for 99mTc-PSMA-I&S radioguided surgery will be determined by the tumor-to-background uptake ratio (TBR) using the time-activity curve function | time from injection to imaging (range: 1-46 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States